CLINICAL TRIAL: NCT05704296
Title: Comparison Between the Saphenous Vein as Y-composite Graft Based on the Left Internal Thoracic Artery Versus Aortocoronary Conduit for Coronary Artery Bypass Grafting: A Prospective Randomized Controlled Trial
Brief Title: Saphenous Vein as Y-composite Versus Aortocoronary Conduit for CABG
Acronym: CONFIG2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ho Young Hwang (Other)
Responsible Party: Sponsor-Investigator, Ho Young Hwang, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2211-023-1376
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery bypass grafting; saphenous vein; coronary angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Saphenous vein as Y-composite graft based on the left internal thoracic artery versus aortocoronary conduit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Y-composite grafting (Experimental): The saphenous vein is anastomosed to the middle portion of the left internal thoracic artery as Y-composite fashion. Then, left anterior descending artery, if targeted, is bypassed with left internal thoracic artery. Other native coronary arterial targets are bypassed with saphenous vein graft.
  Interventions: Procedure: Y-composite grafting
- Aortocoronary grafting (Active Comparator): The saphenous vein is anastomosed to the ascending aorta as aortocoronary fashion. Then, left anterior descending artery, if targeted, is bypassed with left internal thoracic artery. Other native coronary arterial targets are bypassed with saphenous vein graft.
  Interventions: Procedure: Aortocoronary grafting

INTERVENTIONS:
Procedure: Y-composite grafting — Saphenous vein is used as a Y-composite graft during coronary artery bypass grafting
  Arms: Y-composite grafting
Procedure: Aortocoronary grafting — Saphenous vein is used as an aortocoronary graft during coronary artery bypass grafting
  Arms: Aortocoronary grafting

SUMMARY:
Left internal thoracic artery (LITA) has been acknowledged as the first graft of choice for coronary artery bypass grafting (CABG). However, it is still not conclusive which one is the best second graft of choice among right internal thoracic artery, radial artery, right gastroepiploic artery, saphenous vein, and etc., as well as its configuration for CABG.

In our institution, saphenous vein has been primarily used for the second graft and we have harvested it with 'No touch technique'. We have been demonstrated the excellent long-term patency of this 'No touch saphenous vein' in many studies. However, it is still unknown which configuration is the better strategy for the saphenous vein as a Y-composite graft based on the left internal thoracic artery versus an aortocoronary conduit. Thus, we aimed to evaluate morphologic change of saphenous vein graft by 1-year intravascular ultrasound (IVUS) study and angiographic patency results between Y-composite graft and aortocoronary conduit.

DETAILED DESCRIPTION:
The enrolled patient underwent routine sternotomy, and left internal thoracic artery (LITA) and saphenous vein (SV) are harvested. After harvest, the patient is randomized to Y-composite group or aortocoronary group.

For Y-composite group, SV is anastomosed to LITA as Y-composite fashion. Then, LITA is anastomosed to left anterior descending artery. SV is anastomosed to the rest of the target vessels with sequential anastomosis technique (e.g. diagonal branch, obtuse marginal branch, posterolateral branch and posterior descending artery).

For aortocoronary group, LITA is anastomosed to left anterior descending artery. Then, SV is anastomosed to ascending aorta using proximal anastomosis assist device without clamping the aorta. SV is anastomosed to the rest of the target vessels with sequential anastomosis technique (e.g. diagonal branch, obtuse marginal branch, posterolateral branch and posteriori descending artery).

At 1-year follow-up, coronary angiography is performed to evaluate the patency of the saphenous vein graft. Clinical outcomes are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* A patient who is going to receive coronary artery bypass grafting
* Older than 19 years
* Coronary artery bypass grafting is going to be performed with left internal thoracic artery and saphenous vein graft

Exclusion Criteria:

* Other concomitant procedures (e.g. valve or aorta surgery) is planned
* Patients with severe comorbidities which limit the life expectancy of them below 1 year (e.g. terminal cancer)
* Patients whose left internal thoracic artery or saphenous vein is not available due to the low quality, severe injury, or absence of the graft
* Patients whose ascending aorta is not suitable to aortocoronary anastomosis (e.g. ascending aorta aneurysm, porcelain aorta)
* Emergency operation
* Patients who have connective tissue disease
* Reoperative coronary artery bypass grafting

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Graft patency | at postoperative 1 year
  Graft patency measured by coronary angiography

SECONDARY OUTCOMES:
All-cause mortality | at postoperative 1 year
  all deaths from any cause
Cardiac death | at postoperative 1 year
  Any death related to cardiac events, including sudden death during follow-up
Target vessel revascularization | at postoperative 1 year
  Intervention performed for the previously bypassed target vessel during follow-up
Reintervention | at postoperative 1 year
  Any coronary intervention performed during follow-up due to the coronary artery disease
Major Adverse Cardiac Events (MACEs) | at postoperative 1 year
  acute myocardial infarction, coronary reintervention, and cardiac death including sudden death during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ho Young Hwang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because it is not allowed by our Institutional Review Board.